CLINICAL TRIAL: NCT06026488
Title: A Real-World Study of Diffuse Large B-Cell Lymphoma (DLBCL) Patients With Different Genetic Subtypes
Brief Title: Real-World Study of DLBCL With Different Genetic Subtypes
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Principal Investigator, Clinical Professor, Ruijin Hospital
Other Study IDs: DLBCL-RWS-01
Record Dates: First submitted 2023-08-17; First posted 2023-09-07 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: DLBCL - Diffuse Large B Cell Lymphoma; Lymphoma
Keywords: lymphoma; DLBCL; Genetic Subtype; real world analysis
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating; Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All enrolled patients: All patient who signed the consent form for participation to the study
  Interventions: Other: Other

INTERVENTIONS:
Other: Other — real world treatment and survival of DLBCL patients in China

SUMMARY:
To collect and evaluate the data of real-world treatment regimen, efficacy, safety and survival information of DLBCL patients with different genetic suptypes

DETAILED DESCRIPTION:
DLBCL is a highly common malignant tumor in Asia. The aim of the study is to observe and explore the clinical information on DLBCL patients with different genetic subtypes and to analyze the clinical characteristics and prognosis of different molecular subtypes of DLBCL. This study is a non-interventional real world, observational study and all registered data are collected from real clinical practice cases. The medical data includes patient demographic, tumor characteristics, laboratory examination, history of treatments, adverse reactions, efficacy results and possible prognostic factors. The results can guide future precision therapy for DLBCL.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed diffuse large B-cell lymphoma (DLBCL)
* Genetic subtype belonging to at least one of the seven subtypes by using next generation sequencing: MCD, BN2, N1, ST2, A53, EZB (MYC+, MYC-) and others
* Fully comprehension and signature of the informed consent form (ICF) for participation

Exclusion Criteria:

* Those who refuse to use reliable methods of contraception during pregnancy, lactation or age-appropriate period
* Severe mental illness
* Patients deemed unsuitable for inclusion by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: DLBCL patients with genetic subtypes belonging to one of the seven subtypes by NGS: MCD, BN2, N1, ST2, A53, EZB (MYC+, MYC-) and others
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | Baseline up to data cut-off (Up to approximately 9 years)
  Progression-free survival (PFS) is defined as the time from the date of first administration to the date of first disease progression or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
ORR | End of treatment visit (6-8 weeks after last dose on Day 1 of Cycle 6 [Cycle length=21 days]
  Objective Remission Rate (ORR) is defined as the proportion of patients with complete remission (CR) and partial remission (PR)
CRR | End of treatment visit (6-8 weeks after last dose on Day 1 of Cycle 6 [Cycle length=21 days]
  Complete Remission Rate (CRR) is defined as the proportion of patients with CR
OS | Baseline up to data cut-off (Up to approximately 9 years)
  Overall survival (OS) refers to the time from receiving the first dose to death from any cause
DOR | Baseline up to data cut-off (Up to approximately 9 years)
  Duration Of Remission (DOR) refers to the time from the first CR or PR to the time of the first PD or death from any cause
TTR | Approximately up to 1 year
  Time to remission (TTR) refers to the time from recruitment to the time first CR or PR

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China